CLINICAL TRIAL: NCT04953780
Title: 2157GCCC: a Phase I Trial of Calaspargase Pegol-mknl in Combination with High Dose Cytarabine and Idarubicin in Adult Patients with Newly Diagnosed Acute Myeloid Leukemia
Brief Title: 2157GCCC:Phase 1 of Calaspargase Pegol-mknl W/ Cytarabine and Idarubicin in Newly Dx AML
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Ashkan Emadi, MD PHD, Alexander Bland Osborn Endowed Chair and Distinguished Professor of Medical Oncology, West Virginia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2502110131
Record Dates: First submitted 2021-06-15; First posted 2021-07-08 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — calaspargase pegol

STUDY DESIGN:
Intervention Model Description: 4 parallel-arm study of the different dose of Calaspargase Pegol-mknl with combination with High Dose Cytarabine and /or Idarubicin in Adult Patients with Newly Diagnosed Acute Myeloid Leukemia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Calaspargase pegol-mknl dose level 1 (Experimental): Induction Phase (It usually lasts 29 days):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take Idarubicin 12 mg/m2 for three doses in an IV after the first, third, and fifth High-dose Cytarabine.
  * The subject will take a dose of 750 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine every 21 days ( per cycle).
  Consolidation Phase ( One cycle of consolidation lasts 4-8 weeks):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take a dose of 750 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine.
  * A single cycle of consolidation may last between 4-8 weeks in duration.
  Interventions: Drug: Calaspargase pegol-mknl
- Calaspargase pegol-mknl dose level 2 (Experimental): Induction Phase (It usually lasts 29 days):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take Idarubicin 12 mg/m2 for three doses in an IV after the first, third, and fifth High-dose Cytarabine.
  * The subject will take a dose of 1,000 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine every 21 days ( per cycle).
  Consolidation Phase ( One cycle of consolidation lasts 4-8 weeks):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take a dose of 1,000 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine(every 21 days ( per cycle).
  * A single cycle of consolidation may last between 4-8 weeks in duration.
  Interventions: Drug: Calaspargase pegol-mknl
- Calaspargase pegol-mknl dose level 3 (Experimental): Induction Phase (It usually lasts 29 days):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take Idarubicin 12 mg/m2 for three doses in an IV after the first, third, and fifth High- dose Cytarabine.
  * The subject will take a dose of 1,500 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine every 21 days ( per cycle).
  Consolidation Phase ( One cycle of consolidation lasts 4-8 weeks):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take a dose of 1,500 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine.
  * A single cycle of consolidation may last between 4-8 weeks in duration.
  Interventions: Drug: Calaspargase pegol-mknl
- Calaspargase pegol-mknl dose level 4 (Experimental): Induction Phase (It usually lasts 29 days):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take Idarubicin 12 mg/m2 for three doses in an IV after the first, third, and fifth High-dose Cytarabine.
  * The subject will take a dose of 2,000 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine every 21 days ( per cycle).
  Consolidation Phase ( One cycle of consolidation lasts 4-8 weeks):
  * The subject will take Cytarabine 3000 mg/m2 in an IV every 12 hours on days 1, 3, 5 for 6 doses.
  * The subject will take a dose of 2,000 U/m2 of Calaspargase pegol-mknl in an IV after the last (6th) dose of High-dose Cytarabine per cycle.
  * A single cycle of consolidation may last between 4-8 weeks in duration.
  Interventions: Drug: Calaspargase pegol-mknl

INTERVENTIONS:
Drug: Calaspargase pegol-mknl — Calaspargase pegol-mknl

SUMMARY:
Characterizing the regimen limiting toxicity (RLT) of chemotherapeutic drug Calaspargase Pegol-mknl as remission induction and consolidation chemotherapy in patients with newly diagnosed Acute Myeloid Leukemia (AML) and Identifying the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Calaspargase Pegol-mknl.

DETAILED DESCRIPTION:
This is a single center, non-randomized, open-label, phase I study evaluating regimen-limiting toxicities of Calaspargase Pegol-mknl administered intravenously in Adult Patients with Newly Diagnosed Acute Myeloid Leukemia (AML).

The trial will consist of the induction and consolidation phases of therapy. At the induction phase ( it usually lasts for 29 days): a high-dose of Cytarabine will be administered IV for six doses, plus Idarubicin administered IV for three doses and Calaspargase Pegol-mknl administered IV one dose, using a dose-escalation scheme. At the consolidation phase (single cycle of consolidation lasts 4-8 weeks): a high-dose of Cytarabine will be administered IV for six doses, and Calaspargase Pegol-mknl administered IV for one dose, using a dose-escalation scheme.

The FDA (The US Food and Drug Administration) has not approved Calaspargase Pegol-mknl for Adult Patients with Newly Diagnosed Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* A histologically or pathologically confirmed diagnosis of AML based on WHO classification. Patients with myelodysplastic syndromes (MDS) or myeloproliferative neoplasms (MPN) evolving into AML who are candidates for AML induction therapy are eligible for enrollment.
* Age 18-65 years old.
* ECOG performance status < 3.
* Patients must have normal organ function as defined below:

  * Total bilirubin ≤2X the institutional upper limit of normal (ULN) (except in patients with leukemic infiltration of the liver)
  * AST(SGOT)/ALT(SGPT) ≤3X ULN (except if attributable to leukemic infiltration of the liver)
  * Creatinine Clearance (CrCl) ≥ 40 mL/min (except in patients with evidence of tumor lysis syndrome)
  * Left ventricular ejection fraction (LVEF) ≥50%
* Female patients of childbearing potential must have a negative pregnancy test <1 week before enrollment. Female patients of childbearing potential who are sexually active and male patients who are sexually active and have female partners of childbearing potential must agree to use a highly effective method of non-hormonal contraception. Contraception should be used during treatment and for at least 3 months after the last dose of Calaspargase pegol-mknl.
* Ability to understand and willingness to sign a written informed consent document.
* Agree to comply with the study requirements and agrees to come to the clinic/hospital for required study visits

Exclusion Criteria:

* Patients with the following clinical histories are excluded:

  * severe pancreatitis not related to cholelithiasis. Severe acute pancreatitis as defined by lipase elevation >5X ULN and with signs or symptoms
  * unprovoked DVT
  * PE
  * serious or life-threatening thrombosis in any location of the body
  * hemorrhagic or thromboembolic stroke
  * major hemorrhagic event within three weeks before signing ICF; hemorrhage due to thrombocytopenia from underlying AML is excluded
  * patients with hemorrhagic diathesis
  * neurologic/cerebellar disorders that may confound the toxicity monitoring of HiDAC
  * history of serious hypersensitivity reactions to pegylated L-asparaginase therapy
* Patients receiving any other investigational agents or concurrent chemotherapy or immunotherapy. Hydroxyurea for blast count control is permitted before starting treatment and up to a maximum of 10 days after starting treatment on the study.
* Patients with AML with any of the following cytogenetic abnormalities: t(15;17), t(8;21), inv(16), t(16;16).
* Pregnant women and female patients who are lactating and do not agree to stop breast-feeding.
* Uncontrolled undercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled active seizure disorder, or psychiatric illness/social situations that per site Principal Investigator's judgment would limit compliance with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From the first day of treatment until 30 days after receiving Calaspargase Pegol-mknl
  1. Incidence of regimen limiting toxicities (RLTs) and Incidence of treatment-emergent adverse events (TEAE).

SECONDARY OUTCOMES:
1. CR+CRh+CRi | Within 4-8 weeks following completion of induction regimen and completion of consolidation therapy
  Complete remission (CR) + complete remission with partial hematologic recovery (CRh) + complete remission with incomplete count recovery (CRi)
2. The duration of CR/CRh/CRi. | immediately after the intervention
  The duration of Complete remission (CR) / complete remission with partial hematologic recovery (CRh) / complete remission with incomplete count recovery (CRi)
3. Achievement of MRD <0.02% at the end of Induction therapy with Calaspargase pegol-mknl. | During the intervention
  Achievement of MRD <0.02% at the end of Induction therapy with Calaspargase pegol-mknl.
4. Event-free survival (EFS). | From the first date of intervention until the first documented progression or the date of death from any causes, whichever came first, assessed up to 100 months
  Event-free survival (EFS).
5. Overall survival (OS) | From the first date of intervention until the first documented progression or the date of death from any causes, whichever came first, assessed up to 100 months
  Overall survival (OS)
6. Proceeding to allo-HSCT after Calaspargase pegol-mknl treatment | Immediately after the intervention
  Proceeding to allo-HSCT after Calaspargase pegol-mknl treatment
7. Plasma asparagine and glutamine and other amino acids levels at baseline and weekly after administration of Calaspargase pegol-mknl. for four weeks. | At baseline and weekly after administration of Calaspargase pegol-mknl for four weeks
  Plasma asparagine and glutamine and other amino acids levels at baseline and weekly after administration of Calaspargase pegol-mknl. for four weeks.
8.Plasma asparaginase activity at baseline and weekly after administration of Calaspargase pegol-mknl for four weeks | At baseline and weekly after administration of Calaspargase pegol-mknl for four weeks
  Plasma asparaginase activity at baseline and weekly after administration of Calaspargase pegol-mknl for four weeks

OTHER OUTCOMES:
Exploratory Endpoint 1 | After the enrollment of the study subjects
  Measurement of asparagine synthetase mRNA and protein expression in patients who have refractory disease or develop relapse
Exploratory Endpoint 2 | After the enrollment of the study subjects
  Measurement of p90RSK expression and phosphorylation of p70S6K, 4EBP1, and eIF4E in bone marrow cells of Calaspargase pegol-mknl treated patients with AML
Exploratory Endpoint 3 | After the enrollment of the study subjects
  Measurement of protein expression of MCL-1, BCL2 and BCL-XL in bone marrow cells of Calaspargase pegol-mknl treated patients with AML.
Exploratory Endpoint 4 | After the enrollment of the study subjects
  Tissue banking for further molecular and functional testing in the future

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Emadi, MD, PhD, Principal Investigator — West Virginia University
Locations (2):
- United States (2):
  - Greenebaum Cancer Center, University of Maryland Medical Systems, Baltimore, Maryland
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bade NA, Lu C, Patzke CL, Baer MR, Duong VH, Law JY, Lee ST, Sausville EA, Zimrin AB, Duffy AP, Lawson J, Emadi A. Optimizing pegylated asparaginase use: An institutional guideline for dosing, monitoring, and management. J Oncol Pharm Pract. 2020 Jan;26(1):74-92. doi: 10.1177/1078155219838316. Epub 2019 Mar 27. PMID 30917738
- [Background] Freeman SD, Hourigan CS. MRD evaluation of AML in clinical practice: are we there yet? Hematology Am Soc Hematol Educ Program. 2019 Dec 6;2019(1):557-569. doi: 10.1182/hematology.2019000060. PMID 31808906
- [Background] Loken MR, Alonzo TA, Pardo L, Gerbing RB, Raimondi SC, Hirsch BA, Ho PA, Franklin J, Cooper TM, Gamis AS, Meshinchi S. Residual disease detected by multidimensional flow cytometry signifies high relapse risk in patients with de novo acute myeloid leukemia: a report from Children's Oncology Group. Blood. 2012 Aug 23;120(8):1581-8. doi: 10.1182/blood-2012-02-408336. Epub 2012 May 30. PMID 22649108
- [Background] American Cancer Society. Key Statistics for AML. (2020).
- [Background] Lai C, Doucette K, Norsworthy K. Recent drug approvals for acute myeloid leukemia. J Hematol Oncol. 2019 Sep 18;12(1):100. doi: 10.1186/s13045-019-0774-x. PMID 31533852
- [Background] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Background] Emadi A, Zokaee H, Sausville EA. Asparaginase in the treatment of non-ALL hematologic malignancies. Cancer Chemother Pharmacol. 2014 May;73(5):875-83. doi: 10.1007/s00280-014-2402-3. Epub 2014 Feb 11. PMID 24515335
- [Background] Emadi A, Law JY, Strovel ET, Lapidus RG, Jeng LJB, Lee M, Blitzer MG, Carter-Cooper BA, Sewell D, Van Der Merwe I, Philip S, Imran M, Yu SL, Li H, Amrein PC, Duong VH, Sausville EA, Baer MR, Fathi AT, Singh Z, Bentzen SM. Asparaginase Erwinia chrysanthemi effectively depletes plasma glutamine in adult patients with relapsed/refractory acute myeloid leukemia. Cancer Chemother Pharmacol. 2018 Jan;81(1):217-222. doi: 10.1007/s00280-017-3459-6. Epub 2017 Nov 8. PMID 29119293
- [Background] Emadi A. Exploiting AML vulnerability: glutamine dependency. Blood. 2015 Sep 10;126(11):1269-70. doi: 10.1182/blood-2015-07-659508. No abstract available. PMID 26359432
- [Background] Willems L, Jacque N, Jacquel A, Neveux N, Maciel TT, Lambert M, Schmitt A, Poulain L, Green AS, Uzunov M, Kosmider O, Radford-Weiss I, Moura IC, Auberger P, Ifrah N, Bardet V, Chapuis N, Lacombe C, Mayeux P, Tamburini J, Bouscary D. Inhibiting glutamine uptake represents an attractive new strategy for treating acute myeloid leukemia. Blood. 2013 Nov 14;122(20):3521-32. doi: 10.1182/blood-2013-03-493163. Epub 2013 Sep 6. PMID 24014241
- [Background] Capizzi RL, Davis R, Powell B, Cuttner J, Ellison RR, Cooper MR, Dillman R, Major WB, Dupre E, McIntyre OR. Synergy between high-dose cytarabine and asparaginase in the treatment of adults with refractory and relapsed acute myelogenous leukemia--a Cancer and Leukemia Group B Study. J Clin Oncol. 1988 Mar;6(3):499-508. doi: 10.1200/JCO.1988.6.3.499. PMID 3162515
- [Background] Patzke CL, Duffy AP, Duong VH, El Chaer F, Trovato JA, Baer MR, Bentzen SM, Emadi A. Comparison of High-Dose Cytarabine, Mitoxantrone, and Pegaspargase (HAM-pegA) to High-Dose Cytarabine, Mitoxantrone, Cladribine, and Filgrastim (CLAG-M) as First-Line Salvage Cytotoxic Chemotherapy for Relapsed/Refractory Acute Myeloid Leukemia. J Clin Med. 2020 Feb 16;9(2):536. doi: 10.3390/jcm9020536. PMID 32079074
- [Background] Angiolillo AL, Schore RJ, Devidas M, Borowitz MJ, Carroll AJ, Gastier-Foster JM, Heerema NA, Keilani T, Lane AR, Loh ML, Reaman GH, Adamson PC, Wood B, Wood C, Zheng HW, Raetz EA, Winick NJ, Carroll WL, Hunger SP. Pharmacokinetic and pharmacodynamic properties of calaspargase pegol Escherichia coli L-asparaginase in the treatment of patients with acute lymphoblastic leukemia: results from Children's Oncology Group Study AALL07P4. J Clin Oncol. 2014 Dec 1;32(34):3874-82. doi: 10.1200/JCO.2014.55.5763. Epub 2014 Oct 27. PMID 25348002
- [Background] Vrooman LM, Blonquist TM, Stevenson KE, Supko JG, Hunt SK, Cronholm SM, Koch V, Kay-Green S, Athale UH, Clavell LA, Cole PD, Harris MH, Kelly KM, Laverdiere C, Leclerc JM, Michon B, Place AE, Schorin MA, Welch JJG, Neuberg DS, Sallan SE, Silverman LB. Efficacy and Toxicity of Pegaspargase and Calaspargase Pegol in Childhood Acute Lymphoblastic Leukemia: Results of DFCI 11-001. J Clin Oncol. 2021 Nov 1;39(31):3496-3505. doi: 10.1200/JCO.20.03692. Epub 2021 Jul 6. PMID 34228505
- [Background] Li RJ, Jin R, Liu C, Cao X, Manning ML, Di XM, Przepiorka D, Namuswe F, Deisseroth A, Goldberg KB, Blumenthal GM, Pazdur R. FDA Approval Summary: Calaspargase Pegol-mknl For Treatment of Acute Lymphoblastic Leukemia in Children and Young Adults. Clin Cancer Res. 2020 Jan 15;26(2):328-331. doi: 10.1158/1078-0432.CCR-19-1255. Epub 2019 Aug 23. PMID 31444252
- [Background] Li W, Gong X, Sun M, Zhao X, Gong B, Wei H, Mi Y, Wang J. High-dose cytarabine in acute myeloid leukemia treatment: a systematic review and meta-analysis. PLoS One. 2014 Oct 9;9(10):e110153. doi: 10.1371/journal.pone.0110153. eCollection 2014. PMID 25299623
- [Background] Kern W, Estey EH. High-dose cytosine arabinoside in the treatment of acute myeloid leukemia: Review of three randomized trials. Cancer. 2006 Jul 1;107(1):116-24. doi: 10.1002/cncr.21543. PMID 16721819
- [Background] Wetzler M, Andrews C, Ford LA, Tighe S, Barcos M, Sait SN, Block AW, Nowak NJ, Baer MR, Wang ES, Baumann H. Phase 1 study of arsenic trioxide, high-dose cytarabine, and idarubicin to down-regulate constitutive signal transducer and activator of transcription 3 activity in patients aged <60 years with acute myeloid leukemia. Cancer. 2011 Nov 1;117(21):4861-8. doi: 10.1002/cncr.26097. Epub 2011 Mar 31. PMID 21456022
- [Background] Willemze R, Suciu S, Meloni G, Labar B, Marie JP, Halkes CJ, Muus P, Mistrik M, Amadori S, Specchia G, Fabbiano F, Nobile F, Sborgia M, Camera A, Selleslag DL, Lefrere F Sr, Magro D, Sica S, Cantore N, Beksac M, Berneman Z, Thomas X, Melillo L, Guimaraes JE, Leoni P, Luppi M, Mitra ME, Bron D, Fillet G, Marijt EW, Venditti A, Hagemeijer A, Mancini M, Jansen J, Cilloni D, Meert L, Fazi P, Vignetti M, Trisolini SM, Mandelli F, de Witte T. High-dose cytarabine in induction treatment improves the outcome of adult patients younger than age 46 years with acute myeloid leukemia: results of the EORTC-GIMEMA AML-12 trial. J Clin Oncol. 2014 Jan 20;32(3):219-28. doi: 10.1200/JCO.2013.51.8571. Epub 2013 Dec 2. PMID 24297940
- [Background] Weick JK, Kopecky KJ, Appelbaum FR, Head DR, Kingsbury LL, Balcerzak SP, Bickers JN, Hynes HE, Welborn JL, Simon SR, Grever M. A randomized investigation of high-dose versus standard-dose cytosine arabinoside with daunorubicin in patients with previously untreated acute myeloid leukemia: a Southwest Oncology Group study. Blood. 1996 Oct 15;88(8):2841-51. PMID 8874180
- [Background] Bishop JF, Matthews JP, Young GA, Szer J, Gillett A, Joshua D, Bradstock K, Enno A, Wolf MM, Fox R, Cobcroft R, Herrmann R, Van Der Weyden M, Lowenthal RM, Page F, Garson OM, Juneja S. A randomized study of high-dose cytarabine in induction in acute myeloid leukemia. Blood. 1996 Mar 1;87(5):1710-7. PMID 8634416
- [Background] Chien WW, Le Beux C, Rachinel N, Julien M, Lacroix CE, Allas S, Sahakian P, Cornut-Thibaut A, Lionnard L, Kucharczak J, Aouacheria A, Abribat T, Salles G. Differential mechanisms of asparaginase resistance in B-type acute lymphoblastic leukemia and malignant natural killer cell lines. Sci Rep. 2015 Jan 28;5:8068. doi: 10.1038/srep08068. PMID 25626693
- [Background] Hutson RG, Kitoh T, Moraga Amador DA, Cosic S, Schuster SM, Kilberg MS. Amino acid control of asparagine synthetase: relation to asparaginase resistance in human leukemia cells. Am J Physiol. 1997 May;272(5 Pt 1):C1691-9. doi: 10.1152/ajpcell.1997.272.5.C1691. PMID 9176161
- [Background] Richards NG, Kilberg MS. Asparagine synthetase chemotherapy. Annu Rev Biochem. 2006;75:629-54. doi: 10.1146/annurev.biochem.75.103004.142520. PMID 16756505
- [Background] Aslanian AM, Fletcher BS, Kilberg MS. Asparagine synthetase expression alone is sufficient to induce l-asparaginase resistance in MOLT-4 human leukaemia cells. Biochem J. 2001 Jul 1;357(Pt 1):321-8. doi: 10.1042/0264-6021:3570321. PMID 11415466
- [Background] Andrulis IL, Argonza R, Cairney AE. Molecular and genetic characterization of human cell lines resistant to L-asparaginase and albizziin. Somat Cell Mol Genet. 1990 Jan;16(1):59-65. doi: 10.1007/BF01650480. PMID 1968681
- [Background] Aslanian AM, Kilberg MS. Multiple adaptive mechanisms affect asparagine synthetase substrate availability in asparaginase-resistant MOLT-4 human leukaemia cells. Biochem J. 2001 Aug 15;358(Pt 1):59-67. doi: 10.1042/0264-6021:3580059. PMID 11485552
- [Background] Gallinetti J, Harputlugil E, Mitchell JR. Amino acid sensing in dietary-restriction-mediated longevity: roles of signal-transducing kinases GCN2 and TOR. Biochem J. 2013 Jan 1;449(1):1-10. doi: 10.1042/BJ20121098. PMID 23216249
- [Background] Nobukuni T, Joaquin M, Roccio M, Dann SG, Kim SY, Gulati P, Byfield MP, Backer JM, Natt F, Bos JL, Zwartkruis FJ, Thomas G. Amino acids mediate mTOR/raptor signaling through activation of class 3 phosphatidylinositol 3OH-kinase. Proc Natl Acad Sci U S A. 2005 Oct 4;102(40):14238-43. doi: 10.1073/pnas.0506925102. Epub 2005 Sep 21. PMID 16176982
- [Background] Emadi A, Kapadia B, Bollino D, Bhandary B, Baer MR, Niyongere S, Strovel ET, Kaizer H, Chang E, Choi EY, Ma X, Tighe KM, Carter-Cooper B, Moses BS, Civin CI, Mahurkar A, Shetty AC, Gartenhaus RB, Kamangar F, Lapidus RG. Venetoclax and pegcrisantaspase for complex karyotype acute myeloid leukemia. Leukemia. 2021 Jul;35(7):1907-1924. doi: 10.1038/s41375-020-01080-6. Epub 2020 Nov 16. PMID 33199836
- [Background] FDA. CALASPARGASE PEGOL-MKNL FDA approval label <https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/761102s000lbl.pdf> (2018).
- [Background] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Background] Horvath TD, Chan WK, Pontikos MA, Martin LA, Du D, Tan L, Konopleva M, Weinstein JN, Lorenzi PL. Assessment of l-Asparaginase Pharmacodynamics in Mouse Models of Cancer. Metabolites. 2019 Jan 9;9(1):10. doi: 10.3390/metabo9010010. PMID 30634463